CLINICAL TRIAL: NCT02304887
Title: The Relationship Between the Residual Renal Function and Osteoporosis Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Toshihiko Kono (Other)
Responsible Party: Sponsor-Investigator, Toshihiko Kono, Head of Hospital, Tomidahama Hospital
Organization: Tomidahama Hospital (Other)
Other Study IDs: IRB TH No 9-1
Record Dates: First submitted 2014-11-27; First posted 2014-12-02 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-11

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; Bone mineral densisty; Renal function; CKD-MBD
MeSH Terms: conditions — Osteoporosis; Chronic Kidney Disease-Mineral and Bone Disorder | interventions — Denosumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Bisphosphonate
  Interventions: Drug: Bis, SERM Teriparatide, Denosumab
- Selective estrogen receptor modulator
  Interventions: Drug: Bis, SERM Teriparatide, Denosumab
- Teriparatide
  Interventions: Drug: Bis, SERM Teriparatide, Denosumab
- Senosumab
  Interventions: Drug: Bis, SERM Teriparatide, Denosumab

INTERVENTIONS:
Drug: Bis, SERM Teriparatide, Denosumab — Osteoporotic drugs are assigned according to the disease severity, gender, age and so on.

SUMMARY:
The relationship between osteoporosis drugs and kidney damage is unclear. In this study, we plan to reveal relationship between osteoporosis drugs and kidney damage.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD)- mineral and bone disorder (CKD-MBD) is one of the topic in osteoporosis treatment. As many osteoporotic patients are older, many patients are under the deterioration of the renal function. In addition, several drugs might have the potential for kidney damage. But the relationship between osteoporosis drugs and kidney damage is unclear.

The main objective of this study is to reveal relationship between osteoporosis drugs and kidney damage.

ELIGIBILITY:
Inclusion Criteria:

* Osteoporosis patients

Exclusion Criteria:

* eGFR < 15

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Osteoporosis treatment patients
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2006-01; Primary Completion 2018-12 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Longitudinal renal function changes by osteoporotic treatment | Up to 120 months

CONTACTS AND LOCATIONS:
Overall Officials: Rui Niimi, MD, Principal Investigator — Tomidahama Hospital
Locations (1):
- Tomidahama Hospital, Yokkaichi, Mie-ken, Japan